CLINICAL TRIAL: NCT00011258
Title: Paraoxonase and LDL Oxidation in Carotid Artery Disease
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: S006
Record Dates: First submitted 2001-02-14; First posted 2001-02-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-01

CONDITIONS: Carotid Stenosis
Keywords: Atherosclerosis of the carotid arteries; stroke; lipoprotein metabolism; paraoxonase
MeSH Terms: conditions — Carotid Stenosis; Stroke | interventions — Aryldialkylphosphatase

INTERVENTIONS:
Drug: Paraoxonase

SUMMARY:
Atherosclerosis of the carotid arteries is a common cause of stroke. The prevalence and progression of carotid atherosclerosis are believed to be influenced by genetically inherited variations in lipoprotein metabolism. This study investigates the specific role of paraoxonase, an enzyme thought to detoxify atherogenic oxidized low-density lipoprotein. This study compares veterans who have significant carotid atherosclerosis on ultrasound examination with controls without carotid atherosclerosis. Both paraoxonase activity and genotype will be determined and compared between groups. The results may eventually make it possible to screen for a paraoxonase allele that confers high risk of atherosclerosis, and to diminish the risk by early treatment.

DETAILED DESCRIPTION:
Primary Objective:

Atherosclerosis of the carotid arteries is a common cause of stroke. The prevalence and progression of carotid atherosclerosis are believed to be influenced by genetically inherited variations in lipoprotein metabolism. This study investigates the specific role of paraoxonase, an enzyme thought to detoxify atherogenic oxidized low-density lipoprotein. This study compares veterans who have significant carotid atherosclerosis on ultrasound examination with controls without carotid atherosclerosis. Both paraoxonase activity and genotype will be determined and compared between groups. The results may eventually make it possible to screen for a paraoxonase allele that confers high risk of atherosclerosis, and to diminish the risk by early treatment.

Study Abstract:

The general aim of the proposed research is to evaluate the contribution and mechanism of paraoxonase (PON1) genotypic and phenotypic variation (PON1 status) in risk and progression of carotid artery disease (CAAD). We propose to study moderately affected individuals currently being enrolled in a longitudinal, 3-year magnetic resonance imaging (MR) study to evaluate components of MR image as predictors of CAAD progression. We will study the role of PON1 in CAAD progression in this cohort. We will also collect age-, sex-, race-, and hospital- matched controls, to test hypotheses related to the presence or absence of CAAD. We plan to consider the complex genetic architecture of both vascular disease and PON1 effects in vascular disease. In addition to evaluating known paraoxonase (PON1) polymorphisms, we will evaluate PON1 hydrolysis phenotypes. We have shown that these intervening phenotypes can be superior to known genotypes in CAAD prediction. We will also evaluate PON1 polymorphisms that we have recently detected and shown to affect PON1 expression, as well as consider haplotype effects. The specific aims are to: 1) test for PON1 effects in CAAD progression evaluated by 3 year magnetic resonance image follow-up of percent lumen stenosis; 2) test for PON1 effects in moderate CAAD vs. control prediction, including independence of PON1 from traditional cardiovascular risk factors; and 3) evaluate the possible mechanisms of PON1's association with carotid artery disease, specifically PON1's relationship with the susceptibility of LDL to oxidation and variation in LDL density.

Two paraoxonase (PON1) polymorphisms, PON1-Q192R and PON1-L55M have been inconsistently associated with vascular disease. However, plasma PON1 activity phenotypes vary markedly within genotypes. Thus, activity was expected to add to the informativeness of genotype for predicting vascular disease. The case-control study included 212 age and race matched men with mean age 66.4 yr. (range 49-82 yr.); 95% were Caucasian. The 106 carotid artery disease (CAAD) cases had >80% carotid stenosis and the 106 controls had <15% stenosis. Two PON1 substrate hydrolysis rates (paraoxon, POase; diazoxon, DZOase) were significantly lower in cases than in controls and were significant predictors of CAAD using logistic regression (POase, p=0.005, 25% reduced; DZOase, p=0.019, 16% reduced). POase and DZOase were both significant when included in the same model. DZOase predicted vascular disease independently of lipoprotein profile, HDL subfractions, apoAI, and smoking. The marginal effects of PON1-192 (p=0.75) and PON1-55 (p=0.83) genotypes or haplotype (0.70) did not predict case-control status. However, when phenotype was included as a predictor both PON1-192 and PON1-55 genotypes or haplotypes were significant predictors at the 0.05 level. The common methodology of examining PON1-192 and/or PON1-55 genotypes alone may lead to the erroneous conclusion that there is no PON1 role in CAAD. This may have broad implications for the utility of the "genotype only" approach. These results support the benefit of a "level crossing" approach that includes intervening phenotypes in the study of complexly inherited disease

ELIGIBILITY:
Case: Either had a history of surgical carotid endarterectomy or carotid or CT angiogram showing greater than or equal to 80% stenosis in one or more internal carotid artery. Control: An ultrasound documenting internal carotid artery stenosis less than 15% bilaterally.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 1997-03; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States